CLINICAL TRIAL: NCT06335719
Title: Intraoperative Brief Electrical Stimulation to Improve Cross-Face Nerve Grafting Outcomes
Brief Title: Intraoperative Electrical Stimulation to Improve Nerve Grafting Outcome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #22-926
Record Dates: First submitted 2024-03-15; First posted 2024-03-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Facial Paralysis
MeSH Terms: conditions — Facial Paralysis | interventions — BES

STUDY DESIGN:
Intervention Model Description: Patients will undergo all the standard steps of the facial reanimation procedures. The difference in care is 2/3 participants may receive the brief electrical stimulation therapy.
  Other 1/3 of study participants will undergo the surgery as they normally would if they had not chosen to participate.
Who Masked: Participant
Masking Description: This is a randomized, controlled, double-blinded (patient and evaluator) prospective study. Plan is to enroll up to 30 patients, with a minimum of 20 completing full follow-up. Randomization 2:1 treatment to control due to previous peripheral nerve research demonstrating intraoperative stimulation accelerates axonal regeneration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Treatment group undergoes nerve biopsies during surgery. In addition, patients in the treatment group receive brief electrical stimulation therapy for approximately 10 minutes during the first stage cross-face nerve graft surgery.
  Interventions: Procedure: BES
- Control Group (Experimental): Control group undergoes only nerve biopsies during surgery - no brief electrical stimulation.
  Interventions: Procedure: Standard of Care surgery

INTERVENTIONS:
Procedure: BES — Nerve biopsies during surgery + brief electrical stimulation therapy
  Arms: Treatment Group
Procedure: Standard of Care surgery — Nerve biopsies during surgery - no brief electrical stimulation therapy
  Arms: Control Group

SUMMARY:
A research study to find out if brief intraoperative electrical stimulation therapy improves nerve regeneration and smile outcomes following two-stage cross face nerve graft facial reanimation surgery.

DETAILED DESCRIPTION:
Participants that choose to enroll in this study will be randomly assigned in a 2:1 ratio to a "treatment" or "control" group. In either group, patients will receive the same care as they normally would except for two minor differences. First, patients in both groups undergo nerve biopsies during surgery; these biopsies do not affect the length or outcome of surgery. Second, the treatment group will receive brief electrical stimulation therapy for approximately 10 minutes during the first stage cross-face nerve graft surgery.

The purpose of this study is to evaluate efficacy of an intraoperative dose of brief electrical stimulation (BES) to improve axonal regeneration across a cross-face nerve graft (CFNG) using nerve histology and to evaluate clinical outcomes of treatment and control groups using clinician graded, patient reported, and objective smile metric.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-80 years-old with unilateral facial paralysis who are candidates for two- stage CFNG smile reanimation surgery (i.e. CFNG-driven free gracilis muscle transfer (FGMT) or dual innervation FGMT).
2. Agree to participate in the study.

Exclusion Criteria:

1. Bilateral facial paralysis
2. Age less than 18 years-old or older than 80 years-old
3. Comorbid medical condition preventing two-stage CFNG surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate efficacy of an intraoperative dose of brief electrical stimulation (BES) to improve axonal regeneration across a cross-face nerve graft (CFNG) using nerve histology. | 24 months
  Efficacy evaluation

SECONDARY OUTCOMES:
To evaluate clinical outcomes of treatment and control groups using patient reported, and IRB approved CCF Facial Nerve Survey. | 24 months
  Evaluation of Clinical Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Byrne, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No